CLINICAL TRIAL: NCT02739022
Title: Feasibility Trial of the Early Psychological Support for the Critically Ill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lioudmila Karnatovskaia, M.D., Assistant Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-000145
Record Dates: First submitted 2016-03-16; First posted 2016-04-14 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: PICS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Early Psychological Support for the Critically Ill (EPSCI) (Experimental): patients will receive EPSCI in parallel with medical treatment
  Interventions: Behavioral: Early Psychological Support for the Critically Ill (EPSCI)

INTERVENTIONS:
Behavioral: Early Psychological Support for the Critically Ill (EPSCI) — early psychological support based on positive therapeutic suggestion

SUMMARY:
This is a pilot study designed to test feasibility of a psychotherapeutic intervention for the critically ill patients in intensive care units. Intervention is named Early Psychological Support for the Critically Ill (EPSCI)

ELIGIBILITY:
critically ill adults admitted to the medical intensive care unit (ICU) and expected to stay >48 hours

Inclusion criteria:

-mechanically ventilated patients receiving vasopressors

Exclusion criteria:

* history of dementia
* mental retardation
* suicide attempt
* psychotic disorders such as schizophrenia
* patients on comfort care non-English speaking.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Impact of Events Scale-Revised (IES-R) score | 1 year
  rate of PTSD following ICU stay

SECONDARY OUTCOMES:
feasibility of administering Early Psychological Support for the Critically Ill (EPSCI) | 1 year
  how much time therapy takes, how many interruptions, feedback from staff/family/patient
Hospital Anxiety and Depression Scale (HADS) score | 1 year
  rate of anxiety and depression following intensive care unit (ICU) stay
Montreal Cognitive Assessment-Blind (MoCA-blind) score | 1 year
  rate of cognitive dysfunction following ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Lioudmila V Karnatovskaia, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan Y, Gajic O, Schulte PJ, Clark MM, Philbrick KL, Karnatovskaia LV. Feasibility of a Behavioral Intervention to Reduce Psychological Distress in Mechanically Ventilated Patients. Int J Clin Exp Hypn. 2020 Oct-Dec;68(4):419-432. doi: 10.1080/00207144.2020.1795663. Epub 2020 Jul 30. PMID 32730136